CLINICAL TRIAL: NCT06343194
Title: Analysis of Changes in Electromyographic Activity in Aligner Treatment of Adult Patients With and Without Nocturnal Bruxism: Single-centre Interventional Case-control With Device
Brief Title: Changes in Electromyographic Activity in Aligner Treatment of Adult Patients With and Without Nocturnal Bruxism
Acronym: EMG_BRUX
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Waiting agreement for the use of electromiography in the hospital
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6162
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Sleep Bruxism; Masseter Muscle Hypertrophy; Grinding Teeth
Keywords: clear aligners; bruxoff; electromiograph; therapy; masseter muscle contraction; muscle pain
MeSH Terms: conditions — Sleep Bruxism; Masticatory Muscles, Hypertrophy of; Bruxism; Myalgia

STUDY DESIGN:
Intervention Model Description: bruxism patients and non-bruxism patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bruxism patients assessed with Bruxoff ® (Active Comparator): Subjects classified as bruxists based on the diagnostic criteria for sleep bruxism described by the American Academy of Sleeping Medicine, i.e. if they have at least one of the following two points:
  1. The subject reports or is aware of noises of grinding or clamping during sleep.
  2. One or more of the following signs are present:
     * Abnormal wear of teeth;
     * Discomfort, fatigue or pain in the muscles of the face;
     * Hypertrophy of muscles during voluntary clamping;
     * Any abnormalities in the mandibular muscle activity cannot be expressed by other sleep disorders, medical, neurological, drug use or substance abuse;
     * Bruxoff ® cut-off more than 4.
  Interventions: Device: Bruxoff ®
- non-bruxism patients assessed with Bruxoff ® (Active Comparator): Subjects with good health, with no evidence of bruxism symptoms or signs. Bruxoff ® cut-off equal or less than 4.
  Interventions: Device: Bruxoff ®

INTERVENTIONS:
Device: Bruxoff ® — Bruxoff ® is a holter that measures the masseter muscle contraction and heart rate.

SUMMARY:
The purpose of the study is to evaluate the effectiveness of clear aligners on the symptoms and signs reported by bruxism patients.

The aim of the investigators is to evaluate the effect of treatment on the masticatory muscles and the changes related to the tropism of the masseter muscles using Bruxoff ® device, before and after the beginning of the therapy. Bruxoff ® is a holter that assesses the contractions of the masseter muscles and the heart during sleep.

The plan is to compare treatment with clear aligners for bruxism and non-bruxism patients.

The results will allow the investigators to evaluate the progress of clear aligner therapy in bruxism patients and compare them with those of non-bruxism patients.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of the treatment plan with clear aligners;
* Acceptance of informed consent to the study;
* Subjects classified as bruxists based on the diagnostic criteria for sleep bruxism described by the American Academy of Sleeping Medicine.
* Subjects who don't meet the criteria of sleep bruxism by American Academy of Sleeping Medicine in good health.

Exclusion Criteria:

* Patients with morphological and structural alterations to the temporomandibular joint, e.g. Condillary hypertrophy;
* Medical history of neurological diseases, mental disorders and sleep disturbances e.g. restless leg syndrome and insomnia;
* Patients in therapy with myorelaxants or other medicines that affect chewing muscle activity;
* Patients with pacemakers;
* Patients with periodontal diseases;
* Patients with ongoing orthodontic therapy or with prosthetic rehabilitation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in potentials recorded by Bruxoff ® in bruxism patients. | The records with Bruxoff® device are made: before the beginning of the treatment with clear aligner (T0), after 2 months (T1) and after 6 months (T2) from the start of the therapy.
  The primary outcome of the study is the change in potential recorded by Bruxoff®, defined as the variation in nocturnal masseter contraction activity just in bruxism patients treated with aligners.The study aims to evaluate and compare diagnostic records measured with the Bruxoff® at three time points. Each time, the Bruxoff® is used two nights in a row. The purpose of the first night's data collection is to help the patient learn how to apply and use the device to its fullest potential; only the data collected on the second night will be used in the study to determine whether or not the patient has bruxism.
  * The Bruxoff® device is initially administered for two consecutive nights before the start of aligner therapy (T0).
  * 2 months after starting clear aligner therapy (T1), Bruxoff® is given for two consecutive nights.
  * The last 2 records are registered 6 months after the beginning of the treatment with clear aligners (T2).

SECONDARY OUTCOMES:
Change of signs and symptoms of bruxism | The clinical examinations are made: before the beginning of the treatment with clear aligner (T0), after 2 months (T1) and after 6 months (T2) from the start of the therapy.
  The secondary outcome consists in the mutation of signs (i.e. tooth wear) and symptoms (i.e. massetere muscles pain) of bruxism.
  In order to evaluate how occlusal relationships have changed in bruxism patients treated with aligners at the three study times (T0, T1, T2), we compare their clinical condition with non-bruxism patients.
  Furthermore, it's possible to measure the following characteristics during the three study times (T0, T1, and T2), both in the individual group and between patients with and without bruxism, using the Visual Analogue Scale (range 0-10):
  * the mutation of the chewing muscles' pain and of the related migraines;
  * the variation of the functional limitation during routine mandibular movements related to treatment with clear aligners.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cordaro, professor, Principal Investigator — UOC Odontoiatria Generale e Ortodonzia
Locations (1):
- UOC Clinica Odontoiatrica, Policlinico Agostino Gemelli Università Cattolica del Sacro Cuore, Rome, Lazio, Italy

REFERENCES:
- [Background] Lobbezoo F, Naeije M. Bruxism is mainly regulated centrally, not peripherally. J Oral Rehabil. 2001 Dec;28(12):1085-91. doi: 10.1046/j.1365-2842.2001.00839.x. PMID 11874505
- [Background] Ohlmann B, Bomicke W, Behnisch R, Rammelsberg P, Schmitter M. Variability of sleep bruxism-findings from consecutive nights of monitoring. Clin Oral Investig. 2022 Apr;26(4):3459-3466. doi: 10.1007/s00784-021-04314-8. Epub 2021 Dec 3. PMID 34862565
- [Background] Ohlmann B, Rathmann F, Bomicke W, Behnisch R, Rammelsberg P, Schmitter M. Validity of patient self-reports and clinical signs in the assessment of sleep bruxism based on home-recorded electromyographic/electrocardiographic data. J Oral Rehabil. 2022 Jul;49(7):720-728. doi: 10.1111/joor.13327. Epub 2022 Apr 11. PMID 35348247
- [Background] Manfredini D, Ahlberg J, Castroflorio T, Poggio CE, Guarda-Nardini L, Lobbezoo F. Diagnostic accuracy of portable instrumental devices to measure sleep bruxism: a systematic literature review of polysomnographic studies. J Oral Rehabil. 2014 Nov;41(11):836-42. doi: 10.1111/joor.12207. Epub 2014 Jul 8. PMID 25040303
- [Background] Castroflorio T, Bargellini A, Rossini G, Cugliari G, Deregibus A, Manfredini D. Agreement between clinical and portable EMG/ECG diagnosis of sleep bruxism. J Oral Rehabil. 2015 Oct;42(10):759-64. doi: 10.1111/joor.12320. Epub 2015 Jun 7. PMID 26059761
- [Background] Lobbezoo F, Ahlberg J, Glaros AG, Kato T, Koyano K, Lavigne GJ, de Leeuw R, Manfredini D, Svensson P, Winocur E. Bruxism defined and graded: an international consensus. J Oral Rehabil. 2013 Jan;40(1):2-4. doi: 10.1111/joor.12011. Epub 2012 Nov 4. PMID 23121262
- [Background] Lavigne GJ, Huynh N, Kato T, Okura K, Adachi K, Yao D, Sessle B. Genesis of sleep bruxism: motor and autonomic-cardiac interactions. Arch Oral Biol. 2007 Apr;52(4):381-4. doi: 10.1016/j.archoralbio.2006.11.017. Epub 2007 Feb 20. PMID 17313939
- [Background] Bader G, Lavigne G. Sleep bruxism; an overview of an oromandibular sleep movement disorder. REVIEW ARTICLE. Sleep Med Rev. 2000 Feb;4(1):27-43. doi: 10.1053/smrv.1999.0070. PMID 12531159
- [Background] Dube C, Rompre PH, Manzini C, Guitard F, de Grandmont P, Lavigne GJ. Quantitative polygraphic controlled study on efficacy and safety of oral splint devices in tooth-grinding subjects. J Dent Res. 2004 May;83(5):398-403. doi: 10.1177/154405910408300509. PMID 15111632
- [Background] Harada T, Ichiki R, Tsukiyama Y, Koyano K. The effect of oral splint devices on sleep bruxism: a 6-week observation with an ambulatory electromyographic recording device. J Oral Rehabil. 2006 Jul;33(7):482-8. doi: 10.1111/j.1365-2842.2005.01576.x. PMID 16774505
- [Background] Benli M, Ozcan M. Short-term effect of material type and thickness of occlusal splints on maximum bite force and sleep quality in patients with sleep bruxism: a randomized controlled clinical trial. Clin Oral Investig. 2023 Aug;27(8):4313-4322. doi: 10.1007/s00784-023-05049-4. Epub 2023 May 2. PMID 37127807
- [Background] Zheng M, Liu R, Ni Z, Yu Z. Efficiency, effectiveness and treatment stability of clear aligners: A systematic review and meta-analysis. Orthod Craniofac Res. 2017 Aug;20(3):127-133. doi: 10.1111/ocr.12177. Epub 2017 May 26. PMID 28547915
- [Background] Miller KB, McGorray SP, Womack R, Quintero JC, Perelmuter M, Gibson J, Dolan TA, Wheeler TT. A comparison of treatment impacts between Invisalign aligner and fixed appliance therapy during the first week of treatment. Am J Orthod Dentofacial Orthop. 2007 Mar;131(3):302.e1-9. doi: 10.1016/j.ajodo.2006.05.031. PMID 17346581
- [Background] Lou T, Tran J, Castroflorio T, Tassi A, Cioffi I. Evaluation of masticatory muscle response to clear aligner therapy using ambulatory electromyographic recording. Am J Orthod Dentofacial Orthop. 2021 Jan;159(1):e25-e33. doi: 10.1016/j.ajodo.2020.08.012. Epub 2020 Nov 21. PMID 33234460
- [Background] Ciavarella D, Fanelli C, Suriano C, Cazzolla AP, Campobasso A, Guida L, Laurenziello M, Illuzzi G, Tepedino M. Occlusal Plane Modification in Clear Aligners Treatment: Three Dimensional Retrospective Longitudinal Study. Dent J (Basel). 2022 Dec 27;11(1):8. doi: 10.3390/dj11010008. PMID 36661545
- [Background] Bucci R, Rongo R, Levate C, Michelotti A, Barone S, Razionale AV, D'Anto V. Thickness of orthodontic clear aligners after thermoforming and after 10 days of intraoral exposure: a prospective clinical study. Prog Orthod. 2019 Sep 9;20(1):36. doi: 10.1186/s40510-019-0289-6. PMID 31495908
- [Background] Nota A, Caruso S, Ehsani S, Ferrazzano GF, Gatto R, Tecco S. Short-Term Effect of Orthodontic Treatment with Clear Aligners on Pain and sEMG Activity of Masticatory Muscles. Medicina (Kaunas). 2021 Feb 19;57(2):178. doi: 10.3390/medicina57020178. PMID 33669677
- [Background] Yarnitsky D. Conditioned pain modulation (the diffuse noxious inhibitory control-like effect): its relevance for acute and chronic pain states. Curr Opin Anaesthesiol. 2010 Oct;23(5):611-5. doi: 10.1097/ACO.0b013e32833c348b. PMID 20543676
- [Result] Lavigne GJ, Khoury S, Abe S, Yamaguchi T, Raphael K. Bruxism physiology and pathology: an overview for clinicians. J Oral Rehabil. 2008 Jul;35(7):476-94. doi: 10.1111/j.1365-2842.2008.01881.x. PMID 18557915
- [Result] Deregibus A, Castroflorio T, Bargellini A, Debernardi C. Reliability of a portable device for the detection of sleep bruxism. Clin Oral Investig. 2014 Nov;18(8):2037-43. doi: 10.1007/s00784-013-1168-z. Epub 2013 Dec 28. PMID 24374575
- [Result] Kerstein RB, Lowe M, Harty M, Radke J. A force reproduction analysis of two recording sensors of a computerized occlusal analysis system. Cranio. 2006 Jan;24(1):15-24. doi: 10.1179/crn.2006.004. PMID 16541841
- [Result] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Result] Camara-Souza MB, de Figueredo OMC, Rodrigues Garcia RCM. Association of sleep bruxism with oral health-related quality of life and sleep quality. Clin Oral Investig. 2019 Jan;23(1):245-251. doi: 10.1007/s00784-018-2431-0. Epub 2018 Mar 27. PMID 29589157
- [Result] Camara-Souza MB, Figueredo OMC, Rodrigues Garcia RCM. Tongue force, oral health-related quality of life, and sleep index after bruxism management with intraoral devices. J Prosthet Dent. 2020 Oct;124(4):454-460. doi: 10.1016/j.prosdent.2019.07.017. Epub 2019 Dec 9. PMID 31831164
- [Result] Sateia MJ. International classification of sleep disorders-third edition: highlights and modifications. Chest. 2014 Nov;146(5):1387-1394. doi: 10.1378/chest.14-0970. PMID 25367475
- [Result] Saczuk K, Lapinska B, Wilmont P, Pawlak L, Lukomska-Szymanska M. The Bruxoff Device as a Screening Method for Sleep Bruxism in Dental Practice. J Clin Med. 2019 Jun 28;8(7):930. doi: 10.3390/jcm8070930. PMID 31261634
- [Result] Saczuk K, Lapinska B, Wilmont P, Pawlak L, Lukomska-Szymanska M. Relationship between Sleep Bruxism, Perceived Stress, and Coping Strategies. Int J Environ Res Public Health. 2019 Sep 1;16(17):3193. doi: 10.3390/ijerph16173193. PMID 31480550
- [Result] Castroflorio T, Deregibus A, Bargellini A, Debernardi C, Manfredini D. Detection of sleep bruxism: comparison between an electromyographic and electrocardiographic portable holter and polysomnography. J Oral Rehabil. 2014 Mar;41(3):163-9. doi: 10.1111/joor.12131. Epub 2014 Jan 7. PMID 24417585